CLINICAL TRIAL: NCT01340573
Title: Non-Interventional Study Evaluating The Safety and Efficacy In Patients Receiving New PegIntron Pen for Hepatitis C
Brief Title: Evaluating Safety and Efficacy In Hepatitis C Patients After PegIntron Pen Treatment (Study P04896)
Status: Terminated | Type: Observational
Why Stopped: Terminated early due to low enrollment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04896
Record Dates: First submitted 2010-11-18; First posted 2011-04-22 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; pegylated interferon; PegIntron Pen; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Efficacy measurements for sustained viral response HCV RNA were collected at week 24 of study treatment and at week 24 of follow-up in Non-genotype-1 participants. Efficacy measurements for Genotype-1 participants for sustained viral response HCV RNA were collected at week 24 and at week 48 of study treatment, and at week 24 of follow-up.

GROUPS / COHORTS (2):
- Genotype 1 CHC Participants
  Interventions: Drug: PegIntron Pen; Drug: Ribavirin
- Non-genotype 1 CHC participants
  Interventions: Drug: PegIntron Pen; Drug: Ribavirin

INTERVENTIONS:
Drug: PegIntron Pen — Peginterferon alfa-2b, 1.5 microgram/kg each week, administered subcutaneously.
  Other Names: pegylated interferon Pen
Drug: Ribavirin — Dose is based on body weight. Each tablet of ribavirin is 200mg, and given by oral administration. Participants with body weight of <65 kg were administered 800 mg of ribavirin daily, body weight of 65 kg-85 kg received 1000 mg daily, and participants with a body weight of >85 kg received 1200 mg of ribavirin daily.
  Other Names: Ribasphere, Vilona, Copegus, Rebetol, Virazole

SUMMARY:
This is a non-interventional study designed to evaluate the efficacy and safety of combination study drugs in the treatment of participants diagnosed with Chronic Hepatitis C (CHC). CHC participants with confirmed positive hepatitis-C virus (HCV) RNA in plasma, and who have not been previously treated with the Pegylated interferon (PegIntron) Pen, were enrolled into study.

DETAILED DESCRIPTION:
Participants with positive genotype-1 HCV RNA received 48 weeks of treatment of PegIntron Pen plus ribavirin and 24 weeks of follow-up. Participants who were non-genotype-1 HCV RNA positive received 24 weeks of treatment of PegIntron Pen plus ribavirin and 24 weeks of follow-up. Participants were asked to complete a questionnaire to measure the satisfaction and the use of training materials of PegIntron pen using a 1-5 score system provided in the questionnaire. The questionnaire was completed once at first follow-up visit. Efficacy measurements for sustained viral response HCV RNA was collected at week-24 of treatment and at week-24 of follow-up in positive Non-genotype-1 HCV RNA participants. Efficacy measurements for sustained viral response HCV RNA was collected at week-24 and at week-48 of treatment, and at week-24 of follow-up, for positive Genotype-1 HCV RNA participants.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Equal to or greater than 18 years.
* Confirmed chronic hepatitis C with hepatitis C virus (HCV) RNA positive in plasma.
* No previous use of PegIntron Pen.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any interferon or to any of the excipients.
* Pregnant women.
* Women who are breastfeeding.
* Existence of or a history of severe psychiatric condition, particularly severe depression, suicidal ideation or suicide attempt.
* A history of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous six months.
* Severe debilitating medical condition, including patients with chronic renal failure or creatinine clearance < 50 ml/minute.
* Auto immune hepatitis or a history of autoimmune disease.
* Severe hepatic dysfunction or decompensated cirrhosis of the liver.
* Pre-existing thyroid disease unless it can be controlled with conventional treatment.
* Epilepsy and/or compromised central nervous system (CNS) function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indonesian participants ≥18 years of age with confirmed chronic hepatitis C with HCV RNA positive in plasma.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-03-23 (Actual); Primary Completion 2007-10-29 (Actual); Study Completion 2007-10-29 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Genotype 1 CHC Participants and Non-genotype 1 CHC partipants
Period: Overall Study
Arm/Group | All Participants
Started | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  Indonesia | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Genotype-1 Participants Who Experienced Serious Adverse Events (SAE) at Week-48 of Study Treatment
Description: Collection of all safety reports (serious adverse events) from genotype-1 population at week-48 of treatment, from participants on pegylated interferon (PegIntron) pen plus ribavirin.
Time Frame: Week-48
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Genotype-1 Participants Who Experienced Serious Adverse Events (SAE) at Week-24 Follow-up
Description: Collection of all safety reports (serious adverse events) from genotype-1 population at week-24 non-treatment follow-up, from participants on pegylated interferon (PegIntron) pen plus ribavirin.
Time Frame: Week-24 follow-up
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Non-genotype-1 Participants Who Experienced Serious Adverse Events (SAE) at Week-24 of Study Treatment
Description: Collection of all safety reports (serious adverse events) from Non-genotype-1 population at week-24 of study treatment, from participants on pegylated interferon (PegIntron) pen plus ribavirin.
Time Frame: Week-24
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Number of Non-genotype 1 Participants Who Experienced Serious Adverse Events (SAE) on Week-24 Follow-up
Description: Collection of all safety reports (serious adverse events) from Non-genotype-1 population at week-24 non-treatment follow-up, from participants on pegylated interferon (PegIntron) pen plus ribavirin.
Time Frame: Week-24 follow-up
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Non-genotype-1 Participants Who Have Achieved Sustained Virologic Response (SVR) at Week-24 of Study Treatment
Description: Sustained virologic response (SVR) is the absence of detectable HCV RNA in serum after end of treatment.
Time Frame: Week-24
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Non-genotype-1 Participants Who Have Achieved Sustained Virologic Response (SVR) at Week-24 Follow-up
Time Frame: Week-24 follow-up
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Genotype-1 Participants Who Have Achieved Sustained Virologic Response (SVR) at Week-48 of Study Treatment
Time Frame: Week-48
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Genotype-1 Participants Who Have Achieved Sustained Virologic Response (SVR) at Week-24 Follow-up
Time Frame: Week-24 follow-up
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Participants' Overall Rating of Satisfaction and the Use of Training Materials for the Pegintron Pen, as Provided in a Study Questionnaire
Description: Participants will complete a single questionnaire during the first follow-up visit (Week 12). The questionnaire will measure the participant's satisfaction and the use of training materials for the PegIntron Pen during the course of study therapy, as measured by the participant using a 1- 5 score system provided in the questionnaire.
Time Frame: Week 12
Population: The study was terminated early due to low enrollment. This analysis was not performed.
Arm/Group | Genotype 1 CHC Participants | Non-genotype 1 CHC Partipants
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other